CLINICAL TRIAL: NCT03968406
Title: Phase I Study of Talazoparib in Combination With Radiation Therapy for Locally Recurrent Gynecologic Cancers
Brief Title: Talazoparib and Radiation Therapy in Treating Patients With Locally Recurrent Gynecologic Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0899; NCI-2019-00101 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0899 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-02-01; First posted 2019-05-30 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Malignant Female Reproductive System Neoplasm; Recurrent Cervical Carcinoma; Recurrent Endometrial Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Vaginal Carcinoma; Stage IV Cervical Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8; Stage IV Uterine Corpus Cancer AJCC v8; Stage IV Vaginal Cancer AJCC v8; Stage IVA Cervical Cancer AJCC v8; Stage IVA Fallopian Tube Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Primary Peritoneal Cancer AJCC v8; Stage IVA Uterine Corpus Cancer AJCC v8; Stage IVA Vaginal Cancer AJCC v8; Stage IVB Cervical Cancer AJCC v8; Stage IVB Fallopian Tube Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Primary Peritoneal Cancer AJCC v8; Stage IVB Uterine Corpus Cancer AJCC v8; Stage IVB Vaginal Cancer AJCC v8
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Vaginal Neoplasms | interventions — Radiotherapy; Radiation; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (talazoparib, radiation therapy) (Experimental): Patients receive talazoparib PO QD beginning on days -10 to -7 and continuing for up to 8 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy 5 days a week (Monday-Friday) for up to 7 weeks.
  Interventions: Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Talazoparib

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673

SUMMARY:
This phase I trial studies the side effects and best dose of talazoparib in combination with radiation therapy and to see how well they work in treating patients with gynecologic cancers that have come back after previous treatment (recurrent). Talazoparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving talazoparib in combination with radiation therapy may work better in treating patients with gynecologic cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, tolerability, and maximally tolerated dose (MTD) of talazoparib combining talazoparib and fractionated radiotherapy in patients with refractory or recurrent ovarian, fallopian tube, primary peritoneal, cervical, or vaginal or endometrial carcinoma.

SECONDARY OBJECTIVES:

I. To determine the safety profile of talazoparib in combination with fractionated radiotherapy for recurrent gynecologic cancers.

II. To determine a preliminary anti-cancer activity of this combination at the MTD.

EXPLORATORY OBJECTIVES:

I. To explore the potential feasibility of using biomarkers in tumor tissue, whole blood or serum as predictive markers of treatment response.

II. To explore the impact of talazoparib when combined with radiotherapy for recurrent gynecologic cancers on 1) patient reported acute gastrointestinal (GI) toxicity and 2) overall longitudinal quality of life at week 5 of therapy.

OUTLINE: This is a dose escalation study of talazoparib.

Patients receive talazoparib orally (PO) once daily (QD) beginning on days -10 to -7 and continuing for up to 8 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy 5 days a week (Monday-Friday) for up to 7 weeks.

After completion of study treatment, patients are followed up at 1, 3, 6, 9, and 12 months, and then every 6 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Histologically-confirmed recurrent ovarian, fallopian tube, primary peritoneal cancer, endometrial, vaginal, or cervical cancer in the abdomen and pelvis
* Subjects with stage IV disease are eligible as long as disease elsewhere (other than the site(s) to receive radiation therapy [RT]) is undetectable or stable (>= 3 months) and immediate chemotherapy is not required. Willingness to discontinue any cytotoxic chemotherapeutic agents, immunotherapy, biologic therapy, and targeted therapies at least three weeks prior to start of investigational therapy
* Hemoglobin >= 10.0 g/dL and no blood transfusions in the 28 days prior to entry/randomization (choose whichever is most applicable to the study) (within 28 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (within 28 days prior to administration of study treatment)
* No features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) on peripheral blood smear (within 28 days prior to administration of study treatment)
* White blood cells (WBC) > 3 x 10^9/L (within 28 days prior to administration of study treatment)
* Platelet count >= 100 x 10^9/L (within 28 days prior to administration of study treatment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be =< 5 x ULN (within 28 days prior to administration of study treatment)
* Serum creatinine =< 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to administration of study treatment)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1

  * Note: If cannot fulfill ECOG 0-1, must fulfill inclusion criteria below (minimum life expectancy of >= 16 weeks)
* Patients must have a life expectancy >= 16 weeks
* Evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1. Postmenopausal is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments, luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50, radiation-induced oophorectomy with last menses > 1 year ago, chemotherapy-induced menopause with > 1 year interval since last menses, or surgical sterilization (bilateral oophorectomy or hysterectomy)
* Patient of child-bearing potential is willing to adhere to using two forms of highly effective birth control. Condoms with spermicide and one of the following are acceptable: oral contraceptive or hormonal therapy or placement of an intrauterine device (IUD). Acceptable non-hormonal birth control methods include: total sexual abstinence, vasectomized sexual partner plus male condom, tubal occlusion plus male condom with spermicide, IUD plus male condom+spermicide. Acceptable hormonal methods include: etonogestrel implants (i.e. Implanon, Norplan), normal and low dose combined oral pills, norelgestromin/ethinyl estradiol (EE) transdermal system, intravaginal device (i.e. EE and etonogestrel) or cerazette (desogestrel). All of these would need to be combined with male condom with spermicide
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* At least one lesion, not previously irradiated, that can be accurately measured at baseline as >= 10 mm in the longest diameter (except lymph nodes which must have short axis >= 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements
* For inclusion in biomarker endpoint, patients must fulfill the following criterion:

  * Provision of informed consent for tumor biopsies * If a patient declines to participate in tumor biopsies, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study described in this Clinical Study Protocol, so long as they consent to that part

Exclusion Criteria:

* Ascites, peritoneal carcinomatosis, hepatic metastases
* Prior radiotherapy in the region of planned radiotherapy
* Chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within the 3 weeks prior to start of therapy
* Previous enrollment in the present study
* Participation in another clinical study with an investigational product during the last 4 weeks
* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for >= 5 years (will require discussion with study physician)
* Patients receiving any systemic chemotherapy, radiotherapy
* Concomitant use of known CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir
* Concomitant use of known P-gp inhibitors (i.e. dronedarone, quinidine, ranolazine, verapamil, ketoconazole, itraconazole), P-glycoprotein (P-gp) inducers (i.e. rifampin, tipranavir, ritonavir), or breast cancer resistance protein (BCRP) inhibitors (i.e. elacridar [GF120918]) should be avoided. If patients are taking any P-gp inhibitors, P-gp inducers, or BRCP inhibitors, they will need to stop them prior to enrolment on the study
* Persistent toxicities (>= Common Terminology Criteria for Adverse Events [CTCAE] grade 2) with the exception of alopecia, caused by previous cancer therapy
* Resting electrocardiogram (ECG) with corrected QT (QTc) > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
* Patients with myelodysplastic syndrome/acute myeloid leukemia
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 28 days prior to treatment
* Major surgery within 14 days of starting study treatment and patients must have recovered from any effects of any major surgery
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, unstable spinal cord compression (untreated and unstable for at least 28 days prior to study entry), superior vena cava syndrome, extensive bilateral lung disease on high resolution computed tomography (CT) scan or any psychiatric disorder that prohibits obtaining informed consent
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Breast feeding women
* Patients with a known hypersensitivity to talazoparib or any of the excipients of the product
* Patients with uncontrolled seizures
* Patients requiring pelvic and para-aortic radiotherapy (defined as levels L1/T12)
* Patients with isolated vaginal relapse (i.e. no disease in lymph nodes or else where in pelvis/abdomen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 30 days
  MTD is determined by dose limiting toxicity (DLT). The MTD will be determine using the time-to-event Bayesian optimal interval (TITE-BOIN) model, and it is defined as the dose for which the isotonic estimate of the DLT rate is closest to the target DLT rate.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Incidence of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE).
Response rate | From the start of study treatment until documentation of local or regional recurrence, progression, time to next therapy, and death, assessed up to 2 years
  Anti-cancer activity will be measured by response rate by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Each endpoint will be analyzed using the cumulative incidence method when competing events exist or the product-limit method of Kaplan and Meier when competing events are absent. Additionally, competing risk regression or proportional hazards modeling, whichever is appropriate, will be used to examine each endpoint while adjusting for disease. Estimates and 95% intervals will be reported.
Local control rate | From the start of study treatment until documentation of local or regional recurrence, progression, time to next therapy, and death, assessed up to 2 years
  Will be analyzed using the cumulative incidence method when competing events exist or the product-limit method of Kaplan and Meier when competing events are absent. Additionally, competing risk regression or proportional hazards modeling, whichever is appropriate, will be used to examine each endpoint while adjusting for disease. Local control will be summarized as freedom from local failure calculated as 1 minus the cumulative incidence of local or regional recurrence. Estimates and 95% intervals will be reported.
Time to progression | From the start of study treatment until documentation of local or regional recurrence, progression, time to next therapy, and death, assessed up to 2 years
  Will be analyzed using the cumulative incidence method when competing events exist or the product-limit method of Kaplan and Meier when competing events are absent. Additionally, competing risk regression or proportional hazards modeling, whichever is appropriate, will be used to examine each endpoint while adjusting for disease. Estimates and 95% intervals will be reported.
Progression-free survival | From the start of study treatment until documentation of local or regional recurrence, progression, time to next therapy, and death, assessed up to 2 years
  Will be analyzed using the cumulative incidence method when competing events exist or the product-limit method of Kaplan and Meier when competing events are absent. Additionally, competing risk regression or proportional hazards modeling, whichever is appropriate, will be used to examine each endpoint while adjusting for disease. Estimates and 95% intervals will be reported.
Overall survival | From the start of study treatment until documentation of local or regional recurrence, progression, time to next therapy, and death, assessed up to 2 years
  Will be analyzed using the cumulative incidence method when competing events exist or the product-limit method of Kaplan and Meier when competing events are absent. Additionally, competing risk regression or proportional hazards modeling, whichever is appropriate, will be used to examine each endpoint while adjusting for disease. Estimates and 95% intervals will be reported.

OTHER OUTCOMES:
Level of PAR inhibition | Up to 2 years
  Ninety-five percent confidence intervals will be generated for all summary statistics. No formal statistical testing will be completed. Summary statistics and box plots will be created to examine Functional Assessment of Cancer Therapy (FACT) component scores at each assessment time as well as to examine the Expanded Prostate Cancer Index Composite (EPIC) bowel questionnaire measured at week 5. Models will be created to examine impact of dosage upon quality of life (QoL) and acute gastrointestinal (GI) toxicity. In the case of QoL, the models will examine QoL over time using linear mixed models, and we will test for an interaction effect between dose and time to examine whether any potential effects of dose upon QoL change over time. No testing will be completed; 95% confidence intervals will be created for all model coefficients.
Gamma-H2AX and RAD51 foci formation levels | Up to 2 years
  Gamma-H2AX and RAD51 foci formation levels in peripheral mononuclear cells and CTCs will be tested for association with PAR inhibition using Pearson and Spearman correlation methods. An association between germline and tumor BRCA mutation status and PAR inhibition, H2AX. Ninety-five percent confidence intervals will be generated for all summary statistics. No formal statistical testing will be completed.
Functional Assessment of Cancer Therapy (FACT) | Up to 2 years
  Will examine the component scores at each assessment time. as well as to examine the Expanded Prostate Cancer Index Composite (EPIC) bowel questionnaire measured at week 5. . No testing will be completed; 95% confidence intervals will be created for all model coefficients.
Expanded Prostate Cancer Index Composite (EPIC) | Up to 2 years
  Will examine the Expanded Prostate Cancer Index Composite (EPIC) bowel questionnaire measured at week 5. No testing will be completed; 95% confidence intervals will be created for all model coefficients.
Overall quality of life as assessed by the FACT questionnaire | Up to 2 years
  Models will be created to examine impact of dosage upon quality of life (QoL). In the case of QoL, the models will examine QoL over time using linear mixed models, and we will test for an interaction effect between dose and time to examine whether any potential effects of dose upon QoL change over time. No testing will be completed; 95% confidence intervals will be created for all model coefficients.

CONTACTS AND LOCATIONS:
Overall Officials: Lilie L Lin, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org